CLINICAL TRIAL: NCT05589961
Title: Safety and Efficacy of TRPP Therapy in Glioblastoma Multiforme
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HebeiSH_GBM_V1.0
Record Dates: First submitted 2022-09-01; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- integrated treatment regimen(TRPP) (Experimental)
  Interventions: Drug: TMZ

INTERVENTIONS:
Drug: TMZ — After enrollment, temozolomide 50mg/m2 was given orally for QD until progression, and radiotherapy and PF 0.2g/ time for TID were started one week later until progression. Pembrolizumab 200mg once every 3 weeks until progression; The radiotherapy regimen depends on the patient's recurrence and initial treatment.
  Other Names: PD-1; RF

SUMMARY:
The primary objective of this study is to evaluate the safety of an innovative integrated treatment regimen for recurrent glioblastoma , including patients with recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
This study is a single-center, prospective, open-label, single-arm clinical study of an innovative integrated treatment regimen for recurrent glioblastoma multiforme.

The main outcome measurement of the study is to evaluate the safety of the integrated treatment regimen for glioblastoma multiforme. Secondary outcome measurement are OS, PFS, ORR, and quality of life. Safety is evaluated by monitoring adverse events, physical examination results, vital signs, ECG, hematology, and clinical biochemistry. Imaging was performed at the end of every 3 sessions to assess treatment outcome and disease progression. The whole treatment and efficacy will be observed for two years.

ELIGIBILITY:
Inclusion Criteria:

* The pathological result of glioblastoma WHO grade 4;
* Received standard TMZ chemotherapy and radiotherapy;
* It is not suitable to undergo surgical resection of the lesion again or other drug treatment, or the patient refuses other treatment;
* Men and women aged 18-75;
* Disease progression was confirmed by CT or MRI examination within 4 weeks before enrollment;
* KPS score ≥70;
* Expected survival time ≥ 3 months, and can meet the follow-up requirements;
* Within 7 days before the start of treatment, the results of routine blood tests, liver and renal function tests, and hemagglutination laboratory tests meet the following criteria:

Leukocyte (WBC) ≥ 3.0×109/L

Platelets (PLT) ≥ 100×109/L

Neutrophil (ANC) ≥ 1.5×109/L

Hemoglobin (HGB) ≥ 90g/L

Serum albumin ≥2.8g/dL

Aspartate aminotransferase (AST) ≤2.5× upper limit of normal (ULN) (< 5×ULN for liver metastases)

Alanine aminotransferase (ALT) ≤2.5×ULN (≤5×ULN for liver metastases)

Total bilirubin (TIBC) ≤1.5×ULN, patients with liver cancer or liver metastases should ≤2×ULN

Serum creatinine (CR)≤1.5×ULN or creatinine clearance ≥50ml/min

AST and ALT levels ≤ 2.5×ULN, and patients with liver metastases or liver cancer should ≤ 5×ULN

International Normalized ratio (INR) ≤ 1.5

Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN

* Pregnancy should be ruled out for fertile women, and HCG tests for early pregnancy must be negative; Both male and female participants should ensure that they use contraception during the study and continue to use contraception until the end of the follow-up period;
* Volunteer to participate in the clinical study, cooperate with the doctor to carry out the study, and sign the informed consent form.

Exclusion Criteria:

* Participating in another clinical trial;
* Recurrence within 4 weeks after surgery;
* Recurrence within 4 weeks after chemotherapy;
* Recurrence within 4 weeks after radiotherapy;
* Increased intracranial pressure: midline shift ≥5mm, clinically significant visual edema, vomiting and nausea, or poor level of consciousness;
* Have active infection that is not controlled with appropriate anti-infective therapy;
* Patients with mental illness or other conditions, such as uncontrollable heart disease or lung disease, diabetes, etc., cannot comply with the requirements of research treatment and monitoring;
* Organ transplants;
* Pregnant or lactating women; Persons with disabilities (blind, deaf, dumb, mentally disabled, physically disabled) or suffering from mental diseases as prescribed by law; Drug users or patients with a history of adverse drug abuse and alcohol dependence within 5 years;
* Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as a positive hepatitis B surface antigen [HBsAg] test, HBV-DNA ≥ 500 IU/ml and abnormal liver function; Hepatitis C, defined as hepatitis C antibody [HCV-AB] positive, HCV-RNA above the detection limit of the assay, and abnormal liver function) or co-infection with hepatitis B and C;
* Any other factors that the investigator deems inappropriate for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
To Evaluate the Safety of the Integrated Treatment Regimen for Glioblastoma Multiforme | From first dose until 30 days after the last dose (up to approximately 2 years ) (Cycle length= 21 days)
  Evaluating the possible adverse reactions recorded are analyzed, mainly including the number, incidence and severity of radiochemotherapy-related adverse reactions and immune-related adverse reactions (irAE) from the beginning of treatment to the progression of disease.
  Include:
  1. Systemic reaction: such as dizziness, fatigue, bone or muscle pain, etc.;
  2. drug allergic reaction;
  3. Cytopenia caused by myelosuppression may lead to severe infection, bleeding, anemia, etc.;
  4. Gastrointestinal symptoms such as loss of appetite, nausea, vomiting, abdominal pain, diarrhea, constipation, fecal occult blood, gastrointestinal bleeding, etc.;
  5. Immune-related adverse reactions (irAE) : Pneumonia, including immune correlation immunity correlation colitis, correlation immune correlation hepatitis, nephritis, immune related endocrine diseases, immune correlation skin reactions and other immune system Related adverse reactions.

SECONDARY OUTCOMES:
To Evaluate the survival of the Integrated Treatment Regimen for Glioblastoma Multiforme | From first dose until 30 days after the last dose (up to approximately 2 years ) (Cycle length= 63 days)
  Using the RANO criteria as the efficacy evaluation criteria, multimodal MRI and 11C-MET PET/CT examination were performed to distinguish false progression, recurrence and radiation injury if necessary. MDT was discussed when necessary.
  OS:Survival was measured from the start of treatment for 2 years or until death (from any cause within 2 years). Overall survival was estimated by planMeier. Patients who are still alive will be examined at the last contact visit.
  See RANO Standard for specific standards.
To Evaluate the efficacy of the Integrated Treatment Regimen for Glioblastoma Multiforme | From first dose until 30 days after the last dose (up to approximately 2 years ) (Cycle length= 63 days)
  Using the RANO criteria as the efficacy evaluation criteria, multimodal MRI and 11C-MET PET/CT examination were performed to distinguish false progression, recurrence and radiation injury if necessary. MDT was discussed when necessary.
  PFS:Progression-free survival (PFS) was calculated from the date of SD after treatment until the first occurrence of disease progression. Progression-free survival was estimated by Haplan-Meier. Patients who are still alive and have no disease progression will be examined at the last visit/contact. Whether disease progression is due to the primary or metastases should be documented.ORR and quality of life.
  See RANO Standard for specific standards.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Li, Academician, Study Chair — The Second Hospital of Hebei Medical University
Locations (1):
- the Second Hospital of HeBei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No